CLINICAL TRIAL: NCT02763254
Title: A Phase 2 Open Label Study to Investigate the Safety and Clinical Activity of Autologous EBV-specific T Cells (CMD-003) for the Treatment of Patients With EBV Positive Lymphomas
Brief Title: Cellular Immunotherapy for Viral Induced Cancer - EBV Positive Lymphomas
Acronym: CIVIC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient recruitment rate
Sponsor: Cell Medica Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CM-2015-01
Record Dates: First submitted 2016-04-27; First posted 2016-05-05 (Estimated); Results first posted 2019-03-12 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Hodgkin Lymphoma; Lymphoma, Large B-Cell, Diffuse; Post-transplant Lymphoproliferative Disorder
Keywords: Epstein-Barr Virus; DLBCL; PTLD; EBV; CIVIC; HL; T cell
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Large B-Cell, Diffuse; Epstein-Barr Virus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- baltaleucel-T (Experimental): Treatment consist of up to 5 doses of 2x10E7 cells/m2 administered intravenously every 2 weeks.
  Interventions: Biological: baltaleucel-T

INTERVENTIONS:
Biological: baltaleucel-T — Autologous EBV-specific T cells

SUMMARY:
To investigate the efficacy of autologous Epstein-barr virus (EBV)-specific T cells for the treatment of EBV positive Diffuse Large B Cell Lymphoma (DLBCL), Hodgkin Lymphoma (HL) and Post-transplant Lymphoproliferative Disease (PTLD) after failing first line treatment.

ELIGIBILITY:
Inclusion Criteria:

1. The study will include three primary cohorts, with any of the following EBV+ diseases:

   Cohort A - DLBCL, 1) in first or subsequent relapse, not eligible for autologous transplantation following salvage therapy OR 2) relapse following autologous transplantation.

   Cohort B - HL, brentuximab vedotin (BV) treatment failure or unable to tolerate BV.

   Cohort C - PTLD, rituximab treatment failure.
2. Presence of active lymphoma or active PTLD, based on imaging performed within the previous 3 months.
3. Tumor positive for EBV encoded RNA (EBER) based on report from certified laboratory.
4. Absolute lymphocyte count (ALC) >500/µL
5. Male or female ≥ 12 years of age
6. Weight ≥ 35 kg
7. Eastern Cooperative Oncology Group (ECOG) performance score 0-2, inclusively or Lansky score ≥ 60, as age appropriate
8. Able to understand and comply with the requirements of the study and to provide written informed consent or age appropriate assent for pediatric patients.

Exclusion Criteria:

1. Known central nervous system (CNS) lymphoma
2. Primary refractory HL or DLBCL
3. Bulky disease
4. Relapse or progression following previous autologous EBV specific T cell treatment.
5. Use of systemic corticosteroids > 0.5 mg/kg/day prednisolone or equivalent does of alternative corticosteroid within 10 days prior to obtaining 200 mL starting material
6. Positive for HIV, hepatitis B, hepatitis C, syphilis or human T cell leukemia virus (HTLV).
7. Patient is pregnant or lactating
8. Systemic fungal, bacterial, viral or other infection that is not controlled
9. Prior allogeneic hematopoietic stem cell transplantation (allo HSCT)
10. Known history of primary immunodeficiency

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-11; Primary Completion 2018-02-17 (Actual); Study Completion 2018-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Gunter, MD, Study Director — Cell Medica, Inc
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was closed early due to inadequate recruitment.
Period: Overall Study
Arm/Group | Baltaleucel-T
Started | 1
Completed | 0
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Baltaleucel-T
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 1
Cohort B - Hodgkin Lymphoma (HL) [Count of Participants; unit: Participants] — Relapse or refractory HL disease post brentuximab vedotin (BV) or unable to tolerate BV.
  Participants | 1

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response
Description: Best single observed response, complete response (CR) or partial response (PR) per Lugano 2014 Disease Response Criteria, during 12 month follow-up.
Time Frame: 1 year
Population: Subject was withdrawn early before first disease assessment timepoint.
Groups:
- Balteleucel-T: Treatment consist of up to 5 doses of 2x10E7 cells/m2 administered intravenously every 2 weeks.
  balteleucel-T: Autologous EBV-specific T cells
Arm/Group | Balteleucel-T
Number analyzed (Participants) | 0

2. Secondary Outcome: Adverse Events
Description: Adverse events will be recorded from the time of the first investigational cell product dose is administered until 30 days after the last administration. Serious events recorded for up to 1 year after administration.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Balteleucel-T
Number analyzed (Participants) | 1
Participants | 1

ADVERSE EVENTS:
Time Frame: 1 month
Description: Prescheduled hospital admissions, hospital admissions for elective surgery, transfusions, diagnostic procedures are not considered to be SAEs. Events related to progression of the underlying malignancy will likewise not be categorized as serious.
Arm/Group | Baltaleucel-T
All-Cause Mortality (participants affected / at risk) | 1/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baltaleucel-T (N=1)
Cytokine Release Syndrome (Immune system disorders) | 1 (1)
Hemophagocytic Lymphohistiosytosis (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baltaleucel-T (N=1)
Fatigue (General disorders) | 1 (1) — Grade 1
Anemia (Blood and lymphatic system disorders) | 1 (2) — Grade 3
Platelet Count Decreased (Investigations) | 1 (1) — Grade 4

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol (2017-02-21): https://cdn.clinicaltrials.gov/large-docs/54/NCT02763254/Prot_000.pdf